CLINICAL TRIAL: NCT04764045
Title: The Significance of Peripheral Input in Patients With Post Surgery Neuropathic Pain: Evaluation of Trigger Point Anesthesia. A Double-blind, Randomized, Controlled Exploratory Study
Brief Title: The Significance of Peripheral Input
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Finn Borgbjerg Moltke, MD, clinical professor, Bispebjerg Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NP-FM-19
Record Dates: First submitted 2020-03-09; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Neuropathic Pain
Keywords: Peripheral input; Trigger point injection; Post operative pain
MeSH Terms: conditions — Neuralgia; Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine injection in trigger points (Active Comparator): Ropivacaine injection 1 ml in all trigger points in and around scar after operation in knee, shoulder and foot, one time, duration 3 minutes
  Interventions: Drug: Ropivacaine
- Placebo injection in trigger points (Placebo Comparator): Saline injection 1 ml in all trigger points in and around scar after operation in knee, shoulder and foot, one time, duration 3 minutes
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Injection of 1 ml Ropivacaine in all trigger points in and around scar. Injection of 1 ml saline in all trigger points in and around scar.
  Other Names: Saline

SUMMARY:
The investigators want to examine trigger point injections of local anesthetics, in patients with post operative neuropathic pain, determine changes in sensory disturbances such as allodynia, hyperalgesia and thermal sensitivity and examine whether trigger point injections will attenuate pain in rest and activity.

DETAILED DESCRIPTION:
The presence of cutaneous trigger points in the surgical incision of patients with post-surgery pain has been shown in our pain clinic, all patients have persistent pain for more than 3 month and different sensory disturbances.

Examinations with trigger point injections of local anesthetics have been used to determine the influence of peripheral changes and the significance of afferent input on persistent post-surgery neuropathic pain.

In the present study the investigators will document the influence of cutaneous trigger point injections for both subjective pain experience and objective findings in the area such as allodynia, hyperalgesia and thermal sensitivity. The investigators expect reduction in spontaneous pain intensity and de-crease in peripheral sensory disturbances and will determine the significance of peripheral input in persistent neuropathic pain.

The investigators aim to investigate whether injection of local anesthesia into trigger points compared with placebo (saline) injection will attenuate pain and normalize abnormal sensations, such as hyperalgesia and allodynia. The investigators believe this to be an important investigation to understand the mechanisms behind chronic post-surgery pain.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Patients with chronic pain (daily VAS pain scores >30 mm) for at least 3 months after knee, shoulder or foot surgery
* Patients with at least one identifiable trigger point in relation to incision from the knee, shoulder or foot surgery. A trigger point is defined as an ar-ea in relation to the incision from surgery, in which a light pressure from a cotton pin radiate pain to the nearby area, and exudes a motor reflex causing withdrawal of the leg
* A written informed consent to participate in the study after having fully understood the contents of the protocol and restrictions

Exclusion Criteria:

* Patients who cannot cooperate
* Patients who cannot understand or speak Danish.
* Patients with allergy to the drugs used in the study
* Patients in treatment with vitamin K antagonists.
* Patients with other pain conditions
* Patients with diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in worst pain in rest and in activity | 30 minutes
  Change in worst pain assessed on a visual analogue scale (VAS, 0-100 mm) at rest and after stair walking/abduction of shoulder, before and after trigger point injections compared to baseline pain score

SECONDARY OUTCOMES:
Change in area of sensory disturbances | 30 minutes
  Area of pin-prick hyperalgesia, using von Frey filament 60 g and brush allodynia, using Somdic brush, assessed pre- and post-injection. Areas identified at a control day between the two intervention days.
Change in warm and cold detection, threshold and tolerance before and after intervention in area with hyperalgesia compared to normal skin | 30 minutes
  Detection, thresholds and tolerance for cold and heat within the hyperalgesia area compared to normal skin at the contralateral site, before and after trigger point injections. All measures made with Somedic MSA Thermal Stimulator

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wijayasinghe N, Ringsted TK, Bischoff JM, Kehlet H, Werner MU. The role of peripheral afferents in persistent inguinal postherniorrhaphy pain: a randomized, double-blind, placebo-controlled, crossover trial of ultrasound-guided tender point blockade. Br J Anaesth. 2016 Jun;116(6):829-37. doi: 10.1093/bja/aew071. PMID 27199314
- [Background] Haroutounian S, Nikolajsen L, Bendtsen TF, Finnerup NB, Kristensen AD, Hasselstrom JB, Jensen TS. Primary afferent input critical for maintaining spontaneous pain in peripheral neuropathy. Pain. 2014 Jul;155(7):1272-1279. doi: 10.1016/j.pain.2014.03.022. Epub 2014 Apr 2. PMID 24704366
- [Background] Haroutounian S, Ford AL, Frey K, Nikolajsen L, Finnerup NB, Neiner A, Kharasch ED, Karlsson P, Bottros MM. How central is central poststroke pain? The role of afferent input in poststroke neuropathic pain: a prospective, open-label pilot study. Pain. 2018 Jul;159(7):1317-1324. doi: 10.1097/j.pain.0000000000001213. PMID 29570507